CLINICAL TRIAL: NCT05662020
Title: A Parallel-controlled Study to Evaluate the Immunogenicity and Safety of Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli) in Healthy Female Participants Aged 9-26 Years in China
Brief Title: A Study to Evaluate the Immunogenicity and Safety of HPV Vaccine in Healthy Female Participants Aged 9-26 Years in China
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Health Guard Biotechnology, Inc (Industry)
Collaborators: Yunnan Center for Disease Control and Prevention (Other); Mile City Center for Disease Control and Prevention (Unknown); Qiubei County Center for Disease Control and Prevention (Unknown); Yanshan County Center for Disease Control and Prevention (Unknown); National Institutes for Food and Drug Control, China (Other); Shanghai Stem Pharmaceutical Development Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KLWS-V502-04
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Human Papillomavirus Infection
Keywords: CIN; VIN; VaIN; AIN; Cervical cancer; Vaginal cancer; Vulvar cancer; Anal cancer, genital warts; Genital warts
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Anus Neoplasms; Condylomata Acuminata | interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Intervention Model Description: A total of 2,750 participants were enrolled in this study: 9-14 years (2 doses) group was administrated with investigational vaccine on 0 Day, 6th month, and 9-19 years (3 doses) group was administrated with investigational vaccine on 0 Day, 2nd month and 6th month. Both of these two group are of non-randomized, open label design; 20-26 years (3 doses) group was randomized at a 1: 1 ratio to receive the investigational vaccine or the positive control, respectivelyon 0 Day, 2nd month and 6th month.
Who Masked: Participant, Investigator
Masking Description: The Sponsor, investigators and biostatisticians will remain blinded to subject allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Group of Investigational Vaccine (Experimental): 0.5 mL suspension for injection, each 0.5-mL dose contains approximately 30 mcg of HPV Type 6 L1 protein, 40 mcg of HPV Type 11 L1 protein, 60 mcg of HPV Type 16 L1 protein, 40 mcg of HPV Type 18 L1 protein, 20 mcg of HPV Type 31 L1 protein, 20 mcg of HPV Type 33 L1 protein, 20 mcg of HPV Type 45 L1 protein, 20 mcg of HPV Type 52 L1 protein, and 20 mcg of HPV Type 58 L1 protein.
  Interventions: Biological: Recombinant Nonavalent (types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia coli)
- The Group of Active Control Vaccine (Active Comparator): 0.5-mL suspension for injection, each 0.5-mL dose contains approximately 30 mcg of HPV Type 6 L1 protein, 40 mcg of HPV Type 11 L1 protein, 60 mcg of HPV Type 16 L1 protein, 40 mcg of HPV Type 18 L1 protein, 20 mcg of HPV Type 31 L1 protein, 20 mcg of HPV Type 33 L1 protein, 20 mcg of HPV Type 45 L1 protein, 20 mcg of HPV Type 52 L1 protein, and 20 mcg of HPV Type 58 L1 protein.
  Interventions: Biological: GARDASIL® 9

INTERVENTIONS:
Biological: Recombinant Nonavalent (types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia coli) — 9-19 years group (3 doses) and 20-26 years group (3 doses) will be vaccinated at months 0, 2, 6. 9-14 years group (2 doses) will be vaccinated at months 0, 6.
  Arms: The Group of Investigational Vaccine
Biological: GARDASIL® 9 — 20-26 years possitive control group will be vaccinated at months 0, 2 and 6
  Arms: The Group of Active Control Vaccine

SUMMARY:
The study is to evaluate immune response induced by 9-valent HPV study vaccine is non-inferior to those induced by GARDASIL® 9 administrated with 3-dose schedule in female participants aged 20-26 years in China, if the immune response induced with same conditions in 9-19 age group is non-inferior to 20-26 age group, and if the immune response induced by 9-valent HPV study vaccine administrated with 2-dose schedule in females aged 9-14 years is non-inferior to 3-dose schedule in females aged 20-26 years.

DETAILED DESCRIPTION:
This is a parallel-controlled study. A total of 2,750 participants will be enrolled in this study: 9-14 years (2 doses) group and 9-19 years (3 doses) group are of non-randomized, open label design; 20-26 years (3 doses) group will be randomized and blinded.

9-14 age group and group 9-19 age group will be enrolled in two stages: 20 subjects in 9-19 age group will be enrolled first. After assessing the safety data (including laboratory test data) within 7 days of 1st dose vaccination in these 20 subjects, and if the suspension criteria are not met, the remaining 620 subjects in 9-19 age group and 640 subjects in 9-14 age group will be enrolled subsequently. 20-26 age group will be enrolled directly, with no stage entry requirements. Eligible subjects will be enrolled to received vaccines accordingly. Subjects who have reached menarche will undergo urine pregnancy test prior to each dose of vaccination (on the vaccine day.)

ELIGIBILITY:
Inclusion Criteria：

1. Female participants aged 9-26 years at the time of 1st dose vaccination (9 years ≤ age < 27 years).
2. Participants aged 9-17 years can provide proof of ID for themselves and their legal guardians, and the trustee (if appropriate) can provide proof of delegation and ID; participants aged 18-26 years can provide proof of their legal ID.
3. If the female participant is of childbearing age: she must not be pregnant, must not be breastfeeding, and have negative urine pregnancy test before vaccination (on the day of vaccination); voluntarily agree to use effective contraception within 2 weeks prior to enrollment in the study; have no plans to have children and agrees to use effective contraception from the time of enrollment until 1 month after full vaccination.

   Participants whom have not reached menarche: If menarche occurs between enrollment and 1 month after full vaccination, subjects must agree to use effective contraception until 1 month after full vaccination. [Effective contraceptive measures include: oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, extended-release topical contraceptives, hormonal patches, intrauterine device (IUD), sterilization, abstinence, condoms (male), diaphragm, cervical cap, etc.].
4. The legal guardians or trustees of subjects of 9-17 years voluntarily signed the Informed Consent Form (ICF) with informed consent; Subjects of 9-17 years voluntarily signed the ICF for minors with informed consent; Subjects of 18-26 years voluntarily signed the ICF with informed consent.
5. Participants and/or guardians are able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

1. * Fever (axillary temperature ≥ 37.3°C in participants >14 years and ≥ 37.5°C in participants ≤14 years) within 24 hours prior to the 1st dose of vaccination.
2. Previously vaccinated or have plans to administer other HPV vaccines during the study period.
3. Plans to participate in other clinical studies during the study period or participate in other unfinished clinical trials within three months before participating in this clinical study; have used or plan to use other investigational or unregistered products (drugs or vaccines) within 28 days prior to 1st vaccination of this study vaccine.
4. History of HPV positive, history of cervical lesions (e.g., abnormal cervical cancer screening results, history of abnormal cervical biopsy results, including cervical intraepithelial neoplasia (CIN), cervical low grade squamous intraepithelial lesions (LSIL), adenocarcinoma in situ or cervical cancer), history of HPV infection or abnormal cytology test or history of pelvic radiation therapy.
5. History of anogenital disease associated with HPV infection (e.g., genital warts, vulvar intraepithelial neoplasia (VIN), vaginal intraepithelial neoplasia (VaIN), anal intraepithelial neoplasia and associated carcinoma, etc.); or history of STDs (including syphilis, gonorrhea, genital chlamydia, genital herpes, soft chancre, lymphogranuloma venereum, inguinal sarcoidosis, etc.).
6. Abnormalities of grade 1 or higher in the laboratory tests specified in this protocol, confirmed by clinician to be clinically significant (only applicable to the 20 subjects enrolled first in group B during the 1st stage).
7. Allergy to any component of the study vaccine (including aluminum hydroxide adjuvant, sodium chloride, histidine, polysorbate, etc.) or previous serious adverse events to vaccination; previous history of serious allergy, including anaphylaxis, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrotizing reaction (Arthus reaction), severe urticaria, respiratory distress, angio neuroedema, etc.
8. Participants with an impaired immune system or who have been diagnosed with an innate or acquired immune deficiency such as HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune disease.
9. Epilepsy, excluding febrile convulsions under 2 years of age, or alcoholic epilepsy 3 years prior to abstinence from alcohol, or simple epilepsy not requiring treatment in the past 3 years.
10. Current severe liver or kidney disease, serious cardiovascular disease, diabetes, malignancy, serious infectious disease (e.g., tuberculosis, HIV infection, etc.)
11. Untreated/uncontrolled hypertension (systolic blood pressure > 120 mmHg and/or diastolic blood pressure > 80 mmHg) prior to vaccination for age 9-17 years; untreated/uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg) prior to vaccination for age 18 years and older.
12. Physician-diagnosed coagulation abnormalities (e.g., coagulation factor deficiency, coagulopathies, platelet abnormalities) or clotting disorders
13. Absence of spleen, asplenia, and any condition resulting asplenia or splenectomy.
14. Participant has received immunosuppressive therapy within 1 month prior to vaccination or is scheduled to receive such therapy during the visit from the 1st dose to 30 days after full vaccination; e.g., long-term systemic glucocorticoid therapy (≥2 mg/kg/day for 2 weeks or more, e.g., prednisone or equivalent); topical medications (e.g., ointments, eye drops, inhalers, or nasal sprays) are allowed.
15. Have received immunoglobulin products or blood-related products within 3 months prior to the 1st dose, or plan to use such products during visits between the 1st dose and 30 days after full vaccination.
16. * Acute illness or in acute exacerbation of chronic disease or use of antipyretic, analgesic and antiallergic medications (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) within 3 days prior to vaccination.
17. * Administration of inactivated/recombinant/nucleic acid vaccines, etc. (non-attenuated vaccines) within 14 days prior to study entry or attenuated vaccines within 28 days prior to study enrollment.
18. * Participant has donated blood within 1 week prior to enrollment or plans to donate blood during the period of 1st dose vaccination to 30 days after full vaccination.
19. A history of psychiatric disorders or current psychiatric disorders result in the inability to comply with study requirements
20. Based on the judgement of investigator, due to various medical, psychological, social, occupational factors or other conditions that are contrary to the study protocol or could affect the signing of ICF by the subject and/or guardian (trustee).

Criteria for delay of the subsequent doses of vaccination:

Participants with confirmed pregnancy prior to vaccination (on the day of vaccination), should delay vaccination to 6 weeks after termination of pregnancy in addition to having a negative urine pregnancy test.

Vaccination may be delayed after evaluation by the investigator:

1. On the day of vaccination, axillary temperature ≥ 37.3°C measured in participants aged > 14 years; axillary temperature ≥ 37.5°C measured in participants aged ≤ 14 years.
2. Treated with immunomodulators, immunoglobulins, or blood-related products in an interval of less than 3 months with vaccination day.
3. Acute illness or acute exacerbation of a chronic disease or use of antipyretic, analgesic and anti-allergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.) 3 days prior to vaccination.
4. Inadequate interval with other vaccinations (receipt of inactivated/recombinant/nucleic acid vaccine, etc. (non-attenuated vaccine) within 14 days or within 28 days for attenuated vaccine before vaccination).
5. The presence of other conditions that the investigator considers to warrant a delay in vaccination.

   -

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2750 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2028-03-23 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies for study vaccine group | 30 days after full immunization
  Geometric mean titer (GMT) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies (pseudo-virus neutralizing assay) 30 days after full vaccination, for participants in study vaccine group: aged 9-14 years (2 doses) group, aged 9-19 years (3 doses) group and aged 20-26 years (3 doses) group.
Seroconversion Rate (SCR) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies for study vaccine group | 30 days after full immunization
  Seroconversion Rate (SCR) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies (pseudo-virus neutralizing assay) 30 days after full vaccination, for participants in study vaccine group: aged 9-14 years (2 doses) group, aged 9-19 years (3 doses) group and aged 20-26 years (3 doses) group

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies for study vaccine group and possitive control group | 30 days after full immunization
  Geometric mean titer (GMT) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies (pseudo-virus neutralizing assay) 30 days after full vaccination, for participants in study vaccine group: 9-14 years (2 doses) group, 9-19 years (3 doses) group, and participants in control vaccine group: 20-26 years (3 doses) group
Seroconversion Rate (SCR) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies for study vaccine group and possitive control group | 30 days after full immunization
  Seroconversion Rate (SCR) of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies (pseudo-virus neutralizing assay) 30 days after full vaccination, for participants in study vaccine group: 9-14 years (2 doses) group, 9-19 years (3 doses) group, and participants in control vaccine group: 20-26 years (3 doses) group
GMT of anti-HPV 6/11/16/18/31/33/45/52/58 specific IgG antibodies for all subjects | 30 days after full immunization
  GMT of anti-HPV 6/11/16/18/31/33/45/52/58 specific IgG antibodies assessed by enzyme-linked immunosorbent assay (ELISA) 30 days after full vaccination for all participants.
SCR of anti-HPV 6/11/16/18/31/33/45/52/58 specific IgG antibodies for all subjects | 30 days after full immunization
  SCR of anti-HPV 6/11/16/18/31/33/45/52/58 specific IgG antibodies assessed by enzyme-linked immunosorbent assay (ELISA) 30 days after full vaccination for all participants.
GMT of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies after first vaccination | From the 12th month to 72nd month after first dose immunization
  GMT of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies (pseudo-virus neutralizing assay) at 12 months, 24 months, 36 months, 48 months, 60 months and 72 months after first vaccination for all participants.
SCR of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies after first vaccination | From the 12th month to 72nd month after first dose immunization
  SCR of anti-HPV type 6/11/16/18/31/33/45/52/58 neutralizing antibodies (pseudo-virus neutralizing assay) at 12 months, 24 months, 36 months, 48 months, 60 months and 72 months after first vaccination for all participants.
Abnormality rate of laboratory test | Day 3 after each dose
  First 20 subjects enrolled in 9-19 years group: abnormality rate of laboratory test on Day 3 after each dose of vaccination.
Follow up 30 minutes observation after injection to collect the Incidence, intensity, and duration of AEs | 30 minutes after each dose
  Follow up 30 minutes observation after injection to collect the Incidence, intensity, and duration of AEs within 30 minutes after each dose of vaccination for all participants
Collect the questionnaires to gather the information related to the Incidence, intensity, and duration of solicited (local and systemic) AEs which within 7 days after each dose | 0-7 days after each dose
  Collect the Safety follow up Dairy Card (questionnaires) to gather the information related to incidence, intensity, and duration of solicited (local and systemic) AEs which within 7 days after each dose of vaccination for all participants
Collect the questionnaires to gather the information related to Incidence, intensity, and duration of unsolicited AEs which within 30 days after each dose | 0-30 days after each dose
  Collect the Safety follow up Dairy Card (questionnaires) to gather the information related to Incidence, intensity, and duration of unsolicited AEs which within 30 days after each dose of vaccination for all participants
Collect the questionnaires to gather the information related to the Incidence, intensity, and duration of SAE | Through study completion, an average of 6 years
  Collect the Safety follow up Dairy Card (questionnaires) to gather the information related to incidence, intensity, and duration of SAE which within 72 months after first vaccination for all participants.
Collect the questionnaires to gather the information related to the Incidence, intensity, and duration of the occurrence of pregnancy events | Through study completion, an average of 6 years
  Collect the Safety follow up Dairy Card (questionnaires) to gather the information related to incidence, intensity, and duration of the occurrence of pregnancy events which within 72 months after first vaccination for all participants

CONTACTS AND LOCATIONS:
Overall Officials: Yongjiang Liu, Bachelor, Study Chair — Beijing Health Guard Biotechnology, Inc
Locations (1):
- Yunnan Center for Disease Prevention and Control, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
No informed consent was obtained to disclose the subject's data and sample test results